CLINICAL TRIAL: NCT00244101
Title: Delivery Room Management of Premature Infants at High Risk of Respiratory Distress Syndrome
Brief Title: Delivery Room Management Trial of Premature Infants at High Risk of Respiratory Distress Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vermont Oxford Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS 03-233
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Prematurity; respiratory distress syndrome; surfactant; nasal continuous positive airway pressure
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Distress Syndrome | interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PS Group (Active Comparator): Intubation, prophylactic surfactant administration shortly after delivery, and subsequent stabilization on ventilator support.
  Interventions: Drug: PS Group
- NCPAP Group (Experimental): Early stabilization on nasal continuous positive airway pressure (NCPAP) with selected intubation and surfactant administration for clinical indications.
  Interventions: Device: NCPAP Group
- ISX Group (Experimental): Intubation, prophylactic surfactant administration shortly after delivery, and rapid extubation to nasal CPAP.
  Interventions: Drug: ISX Group

INTERVENTIONS:
Drug: PS Group — Intubation, prophylactic surfactant administration shortly after delivery, and subsequent stabilization on ventilator support.
  Other Names: Prophylactic Surfactant Group
  Arms: PS Group
Device: NCPAP Group — Early stabilization on nasal continuous positive airway pressure (NCPAP) with selected intubation and surfactant administration for clinical indications.
  Other Names: Nasal CPAP group
  Arms: NCPAP Group
Drug: ISX Group — Intubation, prophylactic surfactant administration shortly after delivery, and rapid extubation to nasal CPAP.
  Other Names: Intubation, Surfactant Administration, Extubation to Nasal CPAP. ENSURE.
  Arms: ISX Group

SUMMARY:
The best mode of delivery room stabilization for premature infants at high risk for respiratory distress syndrome is unknown. The protocol evaluates the impact of three distinct methods of post-delivery stabilization and subsequent early respiratory care on chronic lung disease and survival in premature infants at high risk for respiratory distress syndrome.

DETAILED DESCRIPTION:
The "Delivery room management of premature infants at high risk of respiratory distress syndrome" protocol compares three distinct methods of post-delivery stabilization and subsequent early respiratory care on chronic lung disease and survival in premature infants at high risk of respiratory distress syndrome. The three approaches to post-delivery care include:

1. Intubation, prophylactic surfactant administration shortly after delivery, and subsequent stabilization on ventilator support.
2. Early stabilization on nasal continuous positive airway pressure (NCPAP) with selective intubation and surfactant administration for clinical indications.
3. Intubation, prophylactic surfactant administration shortly after delivery and rapid extubation to nasal CPAP.

The primary null hypothesis for this study is that no difference will be found in chronic lung disease and/or mortality at 36 weeks adjusted age in premature infants at high risk of RDS, depending on the method of post-delivery stabilization.

The study is a randomized, multicenter trial conducted at participating Vermont Oxford Network Centers. Participating centers will demonstrate competency in the use of nasal CPAP by successfully completing a web-based, educational program and utilizing nasal CPAP in a minimum of 20 infants in their NICU.

Infants likely to be delivered to women presenting to a participating Vermont Oxford Network Center at high risk of premature delivery at gestational age 26 + 0 to 29 + 6 weeks will be eligible for inclusion. Specific inclusion criteria that must be met prior to randomization include:

1. imminent delivery
2. no potentially life-threatening congenital anomaly or genetic syndrome
3. no known lung maturity
4. antenatal steroid status known
5. written and informed consent obtained prior to delivery.

Exclusion criteria will include:

1. stillborn infants (Apgar score of 0 at one minute of age) or
2. infants noted to have a potentially life-threatening congenital anomaly or genetic syndrome noted immediately after delivery.

Eligible infants will have consent obtained prior to delivery. They will be stratified into two groups: 26 + 0 to 27 + 6 weeks gestation and 28 + 0 to 29 + 6 weeks gestation. Shortly before delivery, infants will be randomized to one of the three stabilization strategies detailed below:

1. Intubation, prophylactic surfactant administration shortly after delivery, and subsequent stabilization on ventilator support (PS group).
2. Early stabilization on nasal continuous positive airway pressure (NCPAP) with selected intubation and surfactant administration for clinical indications (NCPAP group).
3. Intubation, prophylactic surfactant administration shortly after delivery, and rapid extubation to nasal CPAP (ISX group).

Infants requiring intubation for respiratory failure during this study (in any of the three groups) may be stabilized on either conventional or high-frequency ventilation. Specific criteria regarding target ranges for blood gases and indications for extubation, subsequent surfactant dosing, management of extubation, and criteria for reintubation, are all detailed in the protocol.

The primary outcome measure is chronic lung disease (defined as documented requirement for supplemental oxygen or respiratory support) or mortality at 36 weeks adjusted age. Secondary outcome measures include a variety of clinical outcomes, as well as issues regarding duration of hospital stay and other resource utilization. Long-term outcomes will be measured by a health care questionnaire at two years of age. A sample size of over 895 infants will be required to demonstrate a 25% reduction in the risk of chronic lung disease at 36 weeks adjusted age.

ELIGIBILITY:
Inclusion Criteria:

Infants likely to be delivered to women presenting to a participating Vermont Oxford Network Center at high risk of premature delivery at gestational age 26 + 0 to 29 + 6 weeks will be eligible for inclusion. Specific inclusion criteria that must be met prior to randomization include:

1. Imminent delivery
2. No potentially life-threatening congenital anomaly or genetic syndrome
3. No known lung maturity
4. Antenatal steroid status known
5. Written, informed consent obtained (on admission or prior to delivery).

Exclusion Criteria:

1. Stillborn (Apgar score of 0 at one minute of age)
2. Noted to have a potentially life-threatening congenital anomaly or genetic syndrome noted immediately after delivery.

Ages: 26 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 648 (Actual)
Dates: Start 2003-08; Primary Completion 2009-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger F Soll, MD, Principal Investigator — Vermont Oxford Network; Michael Dunn, MD, Principal Investigator — Sunnybrook and Women's Hospital, Toronto, Ontario, Canada
Locations (1):
- Vermont Oxford Network, Burlington, Vermont, United States

REFERENCES:
- [Result] Dunn MS, Kaempf J, de Klerk A, de Klerk R, Reilly M, Howard D, Ferrelli K, O'Conor J, Soll RF; Vermont Oxford Network DRM Study Group. Randomized trial comparing 3 approaches to the initial respiratory management of preterm neonates. Pediatrics. 2011 Nov;128(5):e1069-76. doi: 10.1542/peds.2010-3848. Epub 2011 Oct 24. PMID 22025591

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PS Group | NCPAP Group | ISX Group
Started | 209 | 223 | 216
Completed | 209 | 223 | 216
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PS Group | NCPAP Group | ISX Group | Total
Number analyzed (Participants) | 209 | 223 | 216 | 648
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 209 | 223 | 216 | 648
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks of gestation] | 28.0 (1.1) | 28.1 (1.3) | 28.1 (1.1) | 28.0 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 99 | 115 | 332
  Male | 91 | 124 | 101 | 316
Region of Enrollment [Number; unit: participants]
  United States | 209 | 223 | 216 | 648

OUTCOME MEASURES:

1. Primary Outcome: Death or Chronic Lung Disease
Time Frame: at 36 weeks postmenstrual age
Population: intention to treat analysis
Measure: Number; unit: participants
Arm/Group | PS Group | NCPAP Group | ISX Group
Number analyzed (Participants) | 209 | 223 | 216
participants | 76 | 68 | 62
Statistical Analysis 1: Comparison: PS Group vs ISX Group; PS group used as standard of care. Relative risk and 95 % CI calculated for PS (reference) versus ISX or NCPAP; Test type: Superiority or Other; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.59 to 1.03]
Statistical Analysis 2: Comparison: PS Group vs NCPAP Group; PS group used as standard of care. Relative risk and 95% CI calculated for PS (reference) versus NCPAP; Test type: Superiority or Other; Risk Ratio (RR) = 0.57, 95% CI 2-sided [0.25 to 1.27]

2. Primary Outcome: Death
Time Frame: 36 weeks adjusted age
Measure: Count of Participants; unit: Participants
Arm/Group | PS Group | NCPAP Group | ISX Group
Number analyzed (Participants) | 209 | 223 | 216
Participants | 15 | 9 | 15
Statistical Analysis 1: Comparison: PS Group vs ISX Group; PS group used as standard of care. Relative risk and 95 % CI calculated for PS (reference) versus ISX; Test type: Superiority or Other; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.49 to 1.94]
Statistical Analysis 2: Comparison: PS Group vs NCPAP Group; PS group used as standard of care. Relative risk and 95% CI calculated for PS (reference) versus NCPAP; Test type: Superiority or Other; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.64 to 1.09]

ADVERSE EVENTS:
Groups:
- Prophylactic Surfactant: Prophylactic surfactant followed by mechanical ventilation
- Surfactant Extubated to nCPAP: prophylactic surfactant with rapid extubation to bubble nCPAP
- NCPAP: initial management with bubble nCPAP and selective surfactant treatment
Arm/Group | Prophylactic Surfactant | Surfactant Extubated to nCPAP | NCPAP
Serious Adverse Events (participants affected / at risk) | 0/209 | 0/216 | 0/223
Other Adverse Events (participants affected / at risk) | 0/209 | 0/216 | 0/223

LIMITATIONS AND CAVEATS:
The study was stopped after recruitment reached 74% of the projected sample size because of difficulties with enrollment. Because this study could not be blinded, there was a possibility of bias influencing the outcomes if providers managing the infants did not follow strict guidelines.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No